CLINICAL TRIAL: NCT05081934
Title: Feasibility, Acceptability and Preliminary Treatment Effects of Adolescent Community Reinforcement Approach, A-CRA, for Youth in Compulsory Institutional Care
Brief Title: Feasibility, Acceptability and Preliminary Treatment Effects of A-CRA for Youth in Compulsory Institutional Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: National Board of Institutional Care, Sweden (Unknown)
Responsible Party: Principal Investigator, Tobias Lundgren, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-02258
Record Dates: First submitted 2021-09-14; First posted 2021-10-18 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2023-10

CONDITIONS: Substance Use Disorders; Criminal Behavior
MeSH Terms: conditions — Substance-Related Disorders; Criminal Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment as usual, TAU (Active Comparator): TAU: Interventions and treatments usually offered and delivered in institutional care. For example, Motivational Interviewing, MI, Cognitive Behavioral Therapy, CBT, Aggression Replacement Therapy, ART or Acceptance and Commitment Therapy, ACT. Further specification of TAU will be made in collaboration with the institutions included in the trial.
  Interventions: Behavioral: TAU
- TAU + A-CRA (Experimental): Behavioral: A-CRA, a 12-14 weekly sessions long behavioral treatment for youth (ages 12-25) suffering from substance use disorder and co-occurring problems, i.e. criminal behavior. The aim is to increase constructive behavior that reduces the need of substances and creates a context where it is rewarding to stay sober. Individual functional analyses, goals and needs guides treatment planning and interventions.
  TAU: interventions and treatments usually offered and delivered in institutional care. For example, Motivational Interviewing, MI, Cognitive Behavioral Therapy, CBT, Aggression Replacement Therapy, ART or Acceptance and Commitment Therapy, ACT. Further specification of TAU will be made in collaboration with the institutions included in the trial.
  Interventions: Behavioral: A-CRA; Behavioral: TAU

INTERVENTIONS:
Behavioral: A-CRA — 12-14 weekly sessions of A-CRA, a behavioral treatment for youth suffering from substance use disorder and co-occurring problems. The average time for a placement within SiS is for boys 5,9 months and for girls 4,5 months. To further adjust A-CRA to the closed institutional care, frequency of sessions may be increased to twice a week. This is to facilitate maintaining of focus in treatment and closely follow treatment progress. Treatment consists of 18 procedures that aim to reduce problematic behaviors and increase constructive behaviors. Example of procedures are functional analysis of substance use behavior, functional analysis of prosocial behavior, increasing prosocial activities, drink/drug refusal, relapse prevention, anger management and caregiver sessions. Procedures are combined and tailored to youth individual goals and needs.
  Arms: TAU + A-CRA
Behavioral: TAU — Standard care is defined as the interventions and treatments adolescents are usually offered and undergo in institutional care. These are Motivational Interviewing, MI, Cognitive Behavioral Therapy, CBT, Aggression Replacement Therapy, ART or Acceptance and Commitment Therapy, ACT. This will be further specified and registered in the initial phase of the study, in collaboration with SiS.

SUMMARY:
Substance abuse and criminal behavior are increasing among adolescents in Sweden. The Swedish National Board of Institutional Care, SiS, provides institutional care on basis of the Swedish laws Care of Young Persons (Special Provisions) Act, LVU, Care of Substance Abusers (Special Provisions) Act, LVM, Secure Youth Care Act, LSU. Treatment is provided at locked youth residential homes. The Adolescent Community Reinforcement Approach, A-CRA, an empirically supported substance use treatment, promotes long-term abstinence, increases social stability and decreases depression and other co-morbid psychiatric problems. However, A-CRA has mostly been delivered and evaluated within outpatient care. It is unclear whether A-CRA is as effective when delivered in compulsory care where many adolescents with severe substance use disorder and criminal behavior receive treatment. This study is the first part of a larger project with the overall objective to evaluate and adjust A-CRA to the compulsory care provided at National Board of Institutional Care (Statens institutionsstyrelse, SiS) for justice-involved youth. The aim of this first part is to examine feasibility, acceptability and preliminary effects of A-CRA when provided in institutional care (SiS). Furthermore, to explore experiences of undergoing and delivering A-CRA in the institutional setting. Data collected from this study will be used for improvement of a coming full scale randomized controlled trial planned for 2022. Expected results are that A-CRA is feasible in the institutional environment, that A-CRA is perceived as helpful and acceptable by therapists and adolescents, that planned procedures are feasible and data collection and recruitment works satisfactorily.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the feasibility, acceptability and preliminary effects of the empirically supported treatment A-CRA when adjusted to, and delivered in, the institutional care of SiS. Furthermore, to increase pro-social behavior/attitudes and psychological flexibility, to improve mental health and to decrease criminal behavior and substance abuse in youth suffering from substance use disorder and/or disruptive behaviors. This study consists of a qualitative and a quantitative part 1) semi-structured interviews with adolescents and therapists involved in treatment to explore experiences 2) a pilot study to evaluate acceptability, feasibility and preliminary effects of A-CRA. Treatment type and dose (number of sessions received and length of sessions) are registered to enable future analyzes. Acceptability (perceived helpfulness and comprehensibility) is measured using a 7-point Likert-scale, ranging from 1 (not at all helpful) to 7 (very helpful).

Adolescents are randomized to either standard care alone or standard care with the addition of A-CRA. Standard care is defined as the interventions and treatments adolescents are usually offered and undergo in institutional care. These are Motivational Interviewing, MI, Cognitive Behavioral Therapy, CBT, Aggression Replacement Therapy, ART or Acceptance and Commitment Therapy, ACT. This will be further specified and registered in the initial phase of the study, in collaboration with SiS. Randomization takes place at the individual level with even allocation to the groups. Quantitative measurements take place before, during and after treatment as well as follow up once a month for six months. Potential adverse events will be collected after treatment completion using open questions.

ELIGIBILITY:
Inclusion Criteria:

* Age 16-21, placed in institutional care (SiS), with substance use disorder and criminal, violent or destructive behavior, willing and able to undergo A-CRA during their placement.
* Ability to read and understand informed consent.

Exclusion Criteria:

* Severe cognitive or psychiatric condition that obstructs ability to provide informed consent or to undergo assessment or interventions.
* Serious somatic condition requiring acute medical attention.

Ages: 16 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Actual)
Dates: Start 2022-02-16 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Attrition | During treatment and at follow up 6 months.
  Attrition defined as participants discontinuing treatment and assessments.
Inclusion rate. | 0 weeks.
  Proportion of youth accepting to participate after being informed about randomization and offered treatment.
Treatment completion. | Immediately after completion.
  Percentage of treatment completers defined as participants who underwent all planned A-CRA modules.

SECONDARY OUTCOMES:
Completed treatment sessions | Registered weekly
  Proportion of treatment sessions completed in TAU + A-CRA compared to TAU.
Length of treatment sessions | Registered after every session
  Average length of treatment sessions in TAU + A-CRA compared to TAU.
Treatment period | 0 weeks to treatment completion.
  Defined as number of weeks from treatment initiation to treatment completion.
Acceptability of treatment | Post treatment.
  Acceptability is measured using a 7-point Likert-scale, ranging from 1 (not at all helpful) to 7 (very helpful).
Depression, anxiety and stress | 0 weeks, 7 weeks, 14 weeks and at follow up 6 months after treatment.
  Depression Anxiety Stress Scale-21 (DASS-21; Antony, Bieling, Cox, Enns, & Swinson, 1998), a self-assessment scale with three subscales.
Pro-social behavior | 0 weeks, 7 weeks, 14 weeks and at follow up 6 months after treatment.
  Prosocial Tendencies Measure (PTM; Carlo & Randall, 2002), a self-assessment scale measuring pro-social behavior in six domains, such as altruistic, emotional, public and private behavior.
Ongoing alcohol/drug cravings | 0 weeks, 7 weeks, 14 weeks and at follow up 6 months after treatment.
  VAS Single Item Craving Question (Reid, Flammino, Starosta, Palamar, & Franck, 2006), a self-assessment VAS-scale ranging from 0 (no craving) to 100 (maximum craving).
Emotion regulation | 0 weeks, 7 weeks, 14 weeks and at follow up 6 months after treatment.
  Difficulties in Emotion Regulation Scale-16 (DERS-16; Bjureberg et al., 2016), a self-assessment scale measuring problems with emotion regulation in five domains, ability to control impulses in when distressed, non-acceptance of negative emotions, goal orientation when distressed, limited access to emotion regulation strategies perceived as effective and emotional clarity. Consists of 16 items, answers on a Likert-scale ranging from 1 (almost never) to 5 (almost always).
Goal directed behavior, engagement in goal behaviors and obstacles to prosocial and healthy behavioral patterns | 0 weeks, 7 weeks, 14 weeks and at follow up 6 months after treatment.
  Bull's-Eye Values Survey (BEVS; Lundgren et al., 2012). Therapist guided. The scale ranges from 0-7 and is illustrated with a physical metaphor of a dartboard.
Psychological flexibility | 0 weeks, 7 weeks, 14 weeks and at follow up 6 months after treatment.
  Avoidance and Fusion Questionnaire Short Version (AFQ-Y8; Livheim et al.,2016) a self-assessment scale measuring psychological flexibility in adolescents. Consists of 8 items.
Negative effects of treatment | 7 weeks, 14 weeks and at follow up 6 months after treatment.
  Negative Effects Questionnaire (NEQ; Rozental, Kottorp, Boettcher, Andersson, & Carlbring, 2016) NEQ-20 investigate participants' negative effects of psychological treatments. Total range is 0-80, with higher values representing a worse outcome.
Level of Service/Case Management Inventory | 0 weeks, 14 weeks and at follow up 6 months after treatment.
  Level of Service/Case Management Inventory (LS/CMI; Andrews, Bonta, & Wormith, 2000) is a clinician administered instrument to evaluate the risks and needs in youthful offenders and is often used to guide case management. Involves antisocial and pro-criminal attitudes.
Alcohol Use Disorders Identification Test | 0 weeks, 14 weeks and at follow up 6 months after treatment.
  13. Alcohol Use Disorders Identification Test (AUDIT; Saunders et al., 1993) a self-assessment scale screening for hazardous drinking and alcohol abuse disorder.
Drug Use Disorders Identification Test | 0 weeks, 14 weeks and at follow up 6 months after treatment.
  14. Drug Use Disorders Identification Test (DUDIT; Berman, Bergman, Palmstierna, & Schlyter, 2005) a self-assessment scale measuring the use and disorder of drugs.

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Lundgren, PhD, Principal Investigator — Centre for Psychiatry Research, Department of Clinical Neuroscience, Karolinska Institutet
Locations (1):
- Centre for Psychiatry Research, Department of Clinical Neuroscience, Karolinska Institutet., Stockholm, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malarstig I, Tyrberg M, Spannargard A, Garke MA, Lundgren T, Alfonsson S. Adolescent community reinforcement approach in secure care for adolescents with substance use and serious norm-violating behaviour: a randomised feasibility trial. BMJ Open. 2026 Feb 9;16(2):e111332. doi: 10.1136/bmjopen-2025-111332. PMID 41663166